CLINICAL TRIAL: NCT06069843
Title: KET-MCI: An Open-label Trial of Single-dose Ketamine Treatment to Improve Depression in Mild Cognitive Impairment
Brief Title: Single-dose Ketamine Treatment to Improve Depression in Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Rachel Fremont, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00160
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Depression; Mild Cognitive Impairment
Keywords: Depression; Mild Cognitive Impairment; Intravenous Ketamine; Cognition; Neuroplasticity; Geriatric Psychiatry
MeSH Terms: conditions — Depression; Cognitive Dysfunction | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Single dose of IV ketamine administered at the standard dose used for depression treatment (0.5 mg/kg)
  Interventions: Drug: IV Ketamine

INTERVENTIONS:
Drug: IV Ketamine — 0.5 mg/kg IV Ketamine

SUMMARY:
Ketamine is a NMDA-receptor antagonist that promotes synapse formation and has been shown to rapidly improve symptoms in depression. Even a single dose of ketamine has been shown to improve depression and cognition with short-term memory, inhibitory control, cognitive flexibility, and processing speed showing improvements within days of treatment. The mechanism behind ketamine's rapid action is not clear but some groups have speculated it may be related to enhanced neuroplasticity, particularly in the frontal areas and the hippocampus. If this mechanism is accurate, ketamine may be especially effective in treating mild cognitive impairment and depression (MCI-D) where changes in the hippocampus and frontal areas have been implicated. Although few studies have been published on the effects of ketamine in older adults, some small pilot studies suggest that ketamine treatment might be effective in improving depression in older adults and relatively safe. There are no studies looking at the effects of ketamine treatment in patients with MCI-D. The research team hypothesize that IV ketamine treatment will be well-tolerated and will improve depression and cognition in patients with MCI-D. The study team will explore the effects of brain imaging abnormalities and amyloid biomarker status on the responsiveness to ketamine. The study team will conduct an open-label pilot study designed to gather data to support an application for a larger NIH-funded study.

DETAILED DESCRIPTION:
Ketamine is a rapid-acting antidepressant thought to work, at least in part, by the enhancement of neural plasticity and the growth of new synapses. A single dose of ketamine has been shown to improve depression and cognition with short-term memory, inhibitory control, cognitive flexibility, and processing speed showing improvements within days of treatment. The mechanism behind ketamine's rapid action is not clear but some groups have speculated it may be related to enhanced neuroplasticity, particularly in the frontal areas and the hippocampus. If this mechanism is accurate, ketamine may be especially effective in treating individuals with mild cognitive impairment and depression (MCI-D) where changes in the hippocampus and frontal areas have been implicated. Although few studies have been published on the effects of ketamine in older adults, they suggest that ketamine treatment might be effective in improving depression in older adults and relatively safe. There are no studies looking at the effects of ketamine treatment in patients with MCI-D. A key hypothesis of this study is that IV ketamine treatment will be well-tolerated and will improve depression and cognition in patients with MCI-D. The effects of brain imaging and activity abnormalities and amyloid biomarker status on the responsiveness to ketamine will be explored. This open-label pilot study is designed to gather data to support an application for a larger NIH-funded study.

This study is an open-label trial to determine the safety and tolerability of a single sub-anesthetic (0.5 mg/kg) intravenous (IV) ketamine treatment in individuals with mild cognitive impairment and depression (MCI-D). As secondary endpoints, whether treatment with a single dose of ketamine may improve mood or cognition in individuals with MCI-D will be examined. In exploratory analyses, whether AD biomarker status has any influence on the effectiveness of ketamine treatment in MCI and brain connectivity changes after ketamine treatment will be examined. The entire study period will be approximately 1 month from start to finish. The study begins with screening followed by a baseline visit. Then there will be a single visit where an infusion of 0.5 mg/kg of IV ketamine will be performed. There will be follow-up visits 1 day, 2 days, 3 days, 7 days, and one month after the infusion. Baseline visit will include questionnaires, blood draw, cognitive evaluation, clinical evaluation, neuroimaging (specifically a non-contrast magnetic resonance image (MRI)), and an optional electroencephalogram (EEG). Follow-ups will include questionnaires, cognitive evaluation, and clinical evaluation. Additionally, blood draw and imaging (MRI) follow-up may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-90
* Able to give consent
* Montgomery Asberg Depression Rating Scale (MADRS) score of ≥20 consistent with at least "moderate depression"
* Clinical diagnosis of mild cognitive impairment or mild Alzheimer's Disease

Exclusion Criteria:

* Serious unstable medical illness
* Uncontrolled hypertension
* Abnormal electrocardiogram
* Renal impairment defined as BUN 20 mg/dl and/or creatinine clearance >1.3
* Current drug or alcohol use disorder
* History of seizures without a clear or resolved etiology
* Lifetime history of schizophrenia, schizoaffective disorder, or bipolar 1 or 2 disorder
* Montreal Cognitive Assessment (MoCA) score <18
* Presence of psychotic symptoms or lifetime psychotic disorder
* Recreational ketamine or phencyclidine use in the last 2 years
* BMI>40
* Serious or imminent suicidal or homicidal risk
* Systolic blood pressure >165 or diastolic blood pressure >95 on infusion day

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number and severity of symptom events as assessed by the Patient Rated Inventory of Side Effects (PRISE) | end of study, at 1 month
  Number of symptom events as assessed by the patient in a self-report measure. PRISE assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other)
Severity of symptom events as assessed by the Patient Rated Inventory of Side Effects (PRISE) | end of study, at 1 month
  Severity of symptom events as assessed by the patient in a self-report measure. PRISE assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other)
Frequency of symptoms measured using PRISE | end of study, at 1 month
  Frequency of observed adverse events as captured by the PRISE; assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other)

SECONDARY OUTCOMES:
Number of Depressive symptoms as assessed with the Montgomery-Asberg Depression Rating Scale (MADRS) | end of study, at 1 month
  The number of depressive symptoms will be assessed using the Montgomery-Asberg Depression Rating Scale (MADRS). The Montgomery Asberg Depression Rating Scale (MADRS-S) has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression)
Level of cognition as assessed with the NIH Toolbox Cognition Battery | end of study, at 1 month
  The NIH Toolbox Cognition Battery (NIHTB-CB) is a 30 minute long cognitive evaluation consisting of 7 tests done via iPad that has been developed to allow for quick and robust measurement of multiple cognitive domains including executive function, memory, language, and processing speed using a series of well-validated assessments. Scoring for the NIH Toolbox Cognition Battery is automated and individuals are assigned a T-score (mean = 50, SD = 10) representing their cognitive performance compared to age, education, gender, and ethnicity-matched peers.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Fremont, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai (Depression and Anxiety Center), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial where participant has consented to have data shared, after de-identification will be shared.
Supporting Information: Study Protocol
Time Frame: Immediately following publication and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals should be directed to Rachel.fremont@mssm.edu, data requestors will need to sign a data access agreement.